CLINICAL TRIAL: NCT03612843
Title: Clinician-Reported and Patient Reported Incidence of Mild and Significant Adverse Events Associated With Dry Needling by Physical Therapists
Brief Title: Adverse Events in Dry Needling
Status: Completed | Type: Observational
Sponsor: Elizabeth Lane (Other)
Collaborators: Brenau University (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Lane, Co-investigator, University of Utah
Organization: University of Utah (Other)
Other Study IDs: UUtah
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Muscle Soreness; Headache; Knee Osteoarthritis; Back Pain; Neck Pain; Needle Stick; Shoulder Pain; Hip Osteoarthritis
Keywords: dry needling; adverse event; physical therapy
MeSH Terms: conditions — Myalgia; Headache; Osteoarthritis, Knee; Back Pain; Neck Pain; Needlestick Injuries; Shoulder Pain; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dry needle: Dry needling is provided as a part of a comprehensive treatment program by a physical therapist. The patient and the therapist will record any adverse events that occur.
  Interventions: Other: Observational dry needle

INTERVENTIONS:
Other: Observational dry needle — No intervention provided by the study. Observation of any adverse events that occur surrounding dry needling by a physical therapist.

SUMMARY:
The purpose of this prospective cohort survey study is to further explore the incidence of adverse events with dry needling by physical therapists - as well as any differences or similarities between patient-reported vs therapist-reported incidence of AEs.

DETAILED DESCRIPTION:
The study design will comprise of an observational study, where practicing clinicians will log data from dry needling sessions and patients will report via online surveys. Clinician logs will be collected weekly via an online REDCap survey . Patients will be instructed to complete an online REDCap survey in the event that an adverse event occurs. Data will be collected for a period of 4 mo.

Descriptive statistics will be used to calculate frequencies of various AE's and rates of occurrence per 100 treatments. Adverse events will be classified on how frequently they occur, ranging from very common (>1/10 treatments) to very rare (<1/10,000 treatments).

The investigators will then examine for differences between patient-reported and clinician-reported incidences and also explore for any correlations between adverse events and other various reported factors.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that receives dry needling as a part of their care by a physical therapist and consents to provide information

Exclusion Criteria:

* Does not receive dry needling or does not consent to provide information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receiving DN as a regular part of their physical therapy care for any diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse event | 1 week
  adverse events are recorded by the patient and therapist

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Benchmark Physical Therapy, Acworth, Georgia
  - Benchmark Physical Therapy, Cartersville, Georgia
  - Benchmark Physical Therapy, Fort Oglethorpe, Georgia
  - Benchmark Physical Therapy, Marietta, Georgia
  - Benchmark Physical Therapy, Roswell, Georgia
  - Benchmark Physical Therapy, Athens, Tennessee
  - Benchmark Physical Therapy, Hixson, Tennessee
  - Benchmark Physical Therapy, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No